CLINICAL TRIAL: NCT02499042
Title: rEduction of oXygen After Cardiac arresT (EXACT): a Pilot Study
Brief Title: rEduction of oXygen After Cardiac arresT: a Pilot Study
Acronym: EXACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Ambulance Victoria (Other Government); SA Ambulance Service (Unknown); Curtin University (Other); Flinders University (Other)
Responsible Party: Principal Investigator, Professor Stephen Bernard, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF14/2953-2014001634
Record Dates: First submitted 2015-07-08; First posted 2015-07-15 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Heart Arrest
Keywords: post-resuscitation; oxygen therapy; out-of-hospital cardiac arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen reduction (Experimental): post-ROSC oxygen reduced to 2L per minute then delivered to maintain oxygen saturation 90-94% to hospital
  Interventions: Drug: Oxygen
- Standard Care (Active Comparator): post-ROSC oxygen maintained ≥10L per minute to hospital
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — oxygen delivery by ETT/ SGA connected to bag/valve/oxygen reservoir

SUMMARY:
This Phase 2 study aims to determine the feasibility of paramedic titration of oxygen delivery in adult patients who have been resuscitated from OHCA.

DETAILED DESCRIPTION:
This Phase 2 study aims to test whether paramedic titration of oxygen is feasible and results in an equivalent number of patients arriving at the ED with a safe oxygen level compared with the current approach of 100% oxygen.

Hypothesis: There is no difference in the proportion of OHCA patients who arrive at the emergency department with oxygen saturation greater than or equal to 90% whether they received an inspired oxygen fraction of 100% achieved by a flow rate of 10 litres per minute compared to a titrated oxygen fraction achieved by a flow rate of 2 litres per minute.

This is a Phase 2, multi-centre, prospective, randomised study to be conducted in Melbourne and Adelaide.

During cardiac arrest, the patient will receive the current standard of care with oxygen delivery (≥10L/min) by ETT/ SGA connected to bag/valve/ oxygen reservoir.

If ROSC is achieved, all the standard post resuscitation treatments will be given as per current ambulance Clinical Practice Guidelines, except for the amount of oxygen delivered.

The initial ventilation post ROSC for two minutes will be 600mL x 10L/ minute with oxygen flow rate ≥10L/min until a satisfactory pulse oximeter trace and reading is achieved.

After the eligibility criteria are met, the patients will be randomised by the opening of an opaque envelope containing a computer generated allocation to either continued oxygen >10L/min or decreased ("titrated") oxygen 2L/min with a target oxygen saturation of 90-94%.

Patients allocated to oxygen >10L minute ("standard care") will continue on this therapy to hospital.

In the 2L/min oxygen group, the oxygen flow will be changed immediately back to >10L/min if:

* The oxygen saturation falls to <90% at any time, or
* Recurrent cardiac arrest occurs, or
* The pulse oximeter trace fails Following any of these events, this high-flow oxygen will continue to hospital. If a patient is extubated or has a SGA removed post randomisation because of improving conscious state, then standard care will be used (i.e. face mask with oxygen ≥10L/min).

For patients with ROSC in whom intubation is planned, ventilation with high-flow oxygen will continue during the intubation process and randomisation will be delayed until 2 minutes after the ETT is confirmed as correctly placed using ETCO2 and the pulse oximeter trace reads ≥95%.

At ED handover, the patient will receive oxygen therapy as determined by the treating emergency medicine physician.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years)
* Out-of-hospital cardiac arrest of presumed cardiac cause
* Initial cardiac rhythm ventricular fibrillation/ ventricular tachycardia ("shockable")
* Unconscious (Glasgow Coma Scale <9)
* In cardiac arrest on ambulance arrival
* Sustained return of spontaneous circulation (>2 minutes)
* Pulse oximeter trace with oxygen saturation measured at ≥95% on bag/ reservoir with oxygen set at ≥10L/min
* Patient is spontaneous breathing or ventilated using bag/valve/oxygen reservoir via endotracheal tube or SGA (i.e. laryngeal mask airway)

Exclusion Criteria:

* Female who is known or suspected to be pregnant
* Dependant on others for activities of daily living (i.e. facilitated care or nursing home residents)
* "Not for Resuscitation" order
* EMS witnessed arrests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
oxygen saturation ≥90% | baseline
  Oxygen saturation measured on arrival at hospital by paramedics

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bernard, MD, Principal Investigator — Monash University / Alfred Hospital
Locations (2):
- Australia (2):
  - SA Ambulance Service, Adelaide, South Australia
  - Ambulance Victoria, Melbourne, Victoria

REFERENCES:
- [Derived] Bray JE, Hein C, Smith K, Stephenson M, Grantham H, Finn J, Stub D, Cameron P, Bernard S; EXACT Investigators. Oxygen titration after resuscitation from out-of-hospital cardiac arrest: A multi-centre, randomised controlled pilot study (the EXACT pilot trial). Resuscitation. 2018 Jul;128:211-215. doi: 10.1016/j.resuscitation.2018.04.019. Epub 2018 Apr 21. PMID 29684433
- See also: The Australian Resuscitation Outcomes Consortium (Aus-ROC) — https://www.ausroc.org.au/